CLINICAL TRIAL: NCT06746038
Title: Evaluation of Extended Wear Hearing Aid for Mild Hearing Loss
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Collaborators: The Woodlands Hearing Center (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRF-469
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-09

CONDITIONS: Sensorineural Hearing Loss
Keywords: extended wear hearing aid
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Intervention Model Description: A single group of participants will be fit with the extended wear hearing devices and will be tested in both the aided and unaided conditions in various tasks. Conditions will be counterbalanced and all participants will experience the same conditions. Conditions will include unaided, aided with pre-calculation A, and aided with pre-calculation B.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Experimental Group (Experimental): Participants who are fit with study Lyric devices and tested on speech intelligibility and effort using two different fitting algorithms
  Interventions: Device: Extended Wear Hearing Aid

INTERVENTIONS:
Device: Extended Wear Hearing Aid — Extended wear hearing aid means that the device is worn 24 hours per day, 7 days a week for months at a time. However, this study will only fit devices on participants for one testing session lasting 2 hours.
  Other Names: Lyric4

SUMMARY:
This study will assess the benefit of extended wear hearing aids for subjective listening effort, compared to the unaided condition, in adults with mild sensorineural hearing loss.

DETAILED DESCRIPTION:
This study will assess the benefit of extended wear hearing aids for subjective listening effort, compared to the unaided condition, in adults with mild sensorineural hearing loss. Participants will be experienced hearing aid users who have previously worn or currently wear extended wear hearing devices. The primary objective will be to assess subjective listening effort, compared to unaided.

ELIGIBILITY:
Inclusion Criteria:

* Meets requirements outlined on Lyric Candidacy Form
* Current Lyric hearing instrument user
* 18 years of age or older at time of enrollment in the study
* Mild sensorineural hearing loss as defined by WHO, 4 frequency PTA of 20-34 dB HL, in the better hearing ear
* Good understanding (read/write/speak) of the English language
* Willingness to comply with all study requirements

Exclusion Criteria:

* Does not meet requirements outlined on Lyric Candidacy Form (see Chapter 9 of the TMF/ISF for SRF-469)
* Difficulty understanding/reading instructions when corrected for vision loss
* Impairments that would restrict participation in any of the evaluations
* Ear health conditions present at baseline that prevent immediate device replacement
* Conditions that would indicate the need for medical referral prior to hearing aid fitting, according to clinic's standard protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
NASA Task Load Index (NASA-TLX) | Day 1 of 1 day study
  A raw score on six demensions (mental demand, physical demand, temporal demand, frustration, effort, performance) on a scale from 1 (low/good) to 20 (high/poor). A higher score indicates higher levels of subjective effort.

SECONDARY OUTCOMES:
AZBio Speech in noise testing | Day 1 of 1 day study
  The percentage of words correctly repeated by the participant when listening to sentences played from a front speaker at a certain dB level, while background noise is presented simultaneously from four corner speakers. A higher percentage indicates better speech understanding in noise.

CONTACTS AND LOCATIONS:
Locations (1):
- The Woodlands Hearing Center, Shenandoah, Texas, United States

IPD SHARING:
Plan to Share IPD: No